CLINICAL TRIAL: NCT00729768
Title: A Phase II/III, Randomized, Open-Label, Active Controlled, Multicenter Trial to Evaluate the Safety and Efficacy of Efalizumab Compared With Cyclosporine, Both in Combination With Mycophenolate Mofetil and Corticosteroids, As an Immunosuppressant Regimen in De Novo Renal Transplantation
Brief Title: A Study to Evaluate Efalizumab Compared With Cyclosporine As an Immunosuppressant Regimen in De Novo Renal Transplantation
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACD4230g
Record Dates: First submitted 2008-08-02; First posted 2008-08-07 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2009-03

CONDITIONS: Kidney Transplantation
Keywords: Renal transplant; Raptiva
MeSH Terms: interventions — Basiliximab; efalizumab; Mycophenolic Acid; Adrenal Cortex Hormones; Cyclosporine

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: basiliximab; Drug: efalizumab; Drug: mycophenolate mofetil; Drug: corticosteroids
- 2 (Active Comparator)
  Interventions: Drug: basiliximab; Drug: mycophenolate mofetil; Drug: corticosteroids; Drug: cyclosporine

INTERVENTIONS:
Drug: basiliximab — 2 intravenous doses
Drug: efalizumab — Subcutaneous repeating dose
  Arms: 1
Drug: mycophenolate mofetil — Oral repeating dose
Drug: corticosteroids — Repeating doses
Drug: cyclosporine — Oral repeating dose
  Arms: 2

SUMMARY:
This is a Phase II/III, randomized, open-label, active-controlled, multicenter trial to evaluate the safety and efficacy of efalizumab compared with cyclosporine (CsA), when both are given in combination with Mycophenolate Mofetil (MMF) and corticosteroids after induction therapy with basiliximab, as an immunosuppressant regimen in de novo renal transplantation. A total of 200 subjects undergoing either living or cadaveric renal transplantation will be randomly assigned 1:1 to receive either efalizumab + MMF + corticosteroids or CsA + MMF + corticosteroids.

ELIGIBILITY:
Key Inclusion Criteria:

* Have signed the informed consent form and the HIPAA patient information form (United States only)
* Are ≥ 18 years of age
* Are a transplant recipient of at least one HLA-mismatch kidney
* For subjects of reproductive potential (men and women), are willing to use effective contraception, unless abstinence is the chosen method

Key Exclusion Criteria:

* Have a history of previous renal transplant
* Have had a PRA > 25% at any time
* Have a history of or evidence of cancer except for basal cell carcinoma that has been excised and cervical carcinoma in situ
* Have a positive T-cell lymphocytotoxic crossmatch with the use of donor lymphocytes and recipient serum
* Have had previous treatment with efalizumab
* Have used any investigational drug within 28 days or 5 half-lives of screening, whichever is longer
* Have a known contraindication to efalizumab
* Have a history of severe allergic or anaphylactic reactions to monoclonal antibodies
* Have had a known allergic reaction or intolerance to any of the following medications: CsA; MMF; Corticosteroids; Basiliximab
* Are allergic to iodinated contrast media that would preclude GFR measurement with iothalamate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Subject and renal allograft survival | 52 weeks

SECONDARY OUTCOMES:
Glomerular filtration rate | 12 and 52 weeks
Change in glomerular filtration rate | 12 weeks to 52 weeks
Transplant renal biopsies | 52 weeks
Change in metabolic/cardiovascular risk factors | 24 weeks and 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.